CLINICAL TRIAL: NCT04195503
Title: Liver Transplantation in Locally- Advanced, Unresectable, Non-Metastatic Intrahepatic Cholangiocarcinoma Treated With Neoadjuvant Systemic Therapy: A Single-centre, Pilot Study
Brief Title: Liver Transplant for Stable, Advanced Intrahepatic Cholangiocarcinoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-5581
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cholangiocarcinoma, Intrahepatic
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liver transplantation (Other): Surgical Intervention - Liver transplantation
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Surgical removal of liver containing tumor(s) and transplantation of new healthy liver graft

SUMMARY:
Diagnosis of intrahepatic cholangiocarcinoma (iCCA) is an increasingly common form of primary liver cancer, but patients with this diagnosis are not currently eligible for LT. This study proposes to offer LT as an option to patients with advanced, unresectable iCCA who demonstrate at least 6 months of disease stability /regression while receiving standard chemotherapy. Patients will be referred and screened for study participation if they have achieved 6 months of disease stability.

They will be worked up for transplant and if eligible, will be listed. Disease must remain controlled while awaiting transplantation. After transplantation, patients will be followed for disease recurrence and overall survival, while receiving standard post-transplantation followup.

DETAILED DESCRIPTION:
Patients treated with standard of care chemotherapy for unresectable, biopsy-proven intrahepatic cholangiocarcinoma, and who demonstrate stability/regression of disease for a minimum of 6 months, may be eligible for study. Following informed consent and screening, eligible patients with a potential live liver donor (an interested, ABO-compatible individual, without obvious contraindications for donation) will be evaluated for transplantation. During this period, patients will continue to receive chemotherapy and imaging at the usual intervals. Once a patient completes the pre-transplant assessments and is deemed "suitable for transplantation" , the living donor's assessments may begin. If the donor is found suitable, a tentative date will be set for the surgeries. Systemic chemotherapy will be stopped approximately 4 weeks before the surgery date.

At that point, the potential recipient will be reimaged (CT scan). Test results, and inclusion and exclusion criteria will be reviewed to ensure the participant remains eligible to proceed to transplant. If these scans reveal any suspicion of tumor infiltration to surrounding tissues, an exploratory laparotomy or endoscopic ultrasound procedure will be scheduled to allow for visual examination and sampling of those tissues. Tissue samples, such as perihilar fat and/or lymph nodes, will be sent to the pathology department for urgent review. If extrahepatic disease is identified, the participant will be excluded from the study and the transplant will not be performed. Any excluded participants will continue to be followed for the study as "drop outs".

Otherwise, the donor and recipient surgeries will be performed in the standard fashion and with the preferred technique of the surgeon. The patient and donor will receive standard of care post-operative care.

Participants (recipients) will be monitored closely for evidence of tumor recurrence with imaging and blood tests. Results of these tests will be collected until completion of the study follow-up period (5-years after LT). In addition to tumor surveillance, liver transplant status will be assessed at each study timepoint (including graft loss, rejection, liver function tests, and details of immunosuppression). The study will also collect details of any biopsies performed, re-hospitalizations and surgical complications

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older, at time of consent
* Eastern Cooperative Oncology Group (ECOG) score : 0 or 1 at all times from study entry to LT
* Able and willing to provide written informed consent.
* Women of child-bearing potential must agree to use adequate birth control
* Histologically-confirmed diagnosis of iCCa
* Disease is deemed unresectable based on tumor location or underlying liver dysfunction
* No vascular invasion, extra-hepatic disease, or lymph node involvement detected on imaging
* Patients must have ≥ 6 months of disease stability or tumor regression on gemcitabine-based therapy. For patients who have progressed to second-line therapy, disease must also be controlled for ≥ 6 months on that regimen
* At least 1 living donor has stepped forward, is blood group compatible and has completed a "Health History form" which, upon review by the Living Donor team, is deemed acceptable and demonstrates no obvious contraindications to donation.

Exclusion Criteria:

* Previous or concurrent cancer (some exceptions permitted)
* Patients who have extrahepatic metastases, lymph node involvement, invasion or encasement of major hepatic vascular structures, perforation of the visceral peritoneum, invasion of extrahepatic structures, invasion of perihilar fat, periductular invasion, concurrent hepatoma or mixed hepatocellular cholangiocarcinoma
* Patients having received prior locoregional therapies or radiation to the tumor
* Renal dysfunction with an estimated creatinine clearance of less than 50 ml/min
* Known history of human immunodeficiency virus (HIV) infection.
* Prior history of solid organ or bone marrow transplantation
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients (unless willing to abstain from breast-feeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
patient survival | 5 years

SECONDARY OUTCOMES:
disease-free survival | 5 years
patient survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lunsford KE, Javle M, Heyne K, Shroff RT, Abdel-Wahab R, Gupta N, Mobley CM, Saharia A, Victor DW, Nguyen DT, Graviss EA, Kaseb AO, McFadden RS, Aloia TA, Conrad C, Li XC, Monsour HP, Gaber AO, Vauthey JN, Ghobrial RM; Methodist-MD Anderson Joint Cholangiocarcinoma Collaborative Committee (MMAJCCC). Liver transplantation for locally advanced intrahepatic cholangiocarcinoma treated with neoadjuvant therapy: a prospective case-series. Lancet Gastroenterol Hepatol. 2018 May;3(5):337-348. doi: 10.1016/S2468-1253(18)30045-1. Epub 2018 Mar 13. PMID 29548617
- [Derived] Achurra P, Fernandes E, O'Kane G, Grant R, Cattral M, Sapisochin G. Liver transplantation for intrahepatic cholangiocarcinoma: who, when and how. Curr Opin Organ Transplant. 2024 Apr 1;29(2):161-171. doi: 10.1097/MOT.0000000000001136. Epub 2024 Jan 23. PMID 38258823